CLINICAL TRIAL: NCT03712319
Title: Mindfulness for Healthcare Students: Smartphone App or Face-to-face Group? A Randomized Controlled Trial
Brief Title: Mindfulness App Versus Mindfulness-based Intervention for Healthcare Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DHAERMP
Record Dates: First submitted 2018-05-25; First posted 2018-10-19 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2018-05

CONDITIONS: Students
Keywords: mindfulness; mobile application; students; anxiety; depression; self-compassion; empathy; burnout
MeSH Terms: conditions — Anxiety Disorders; Depression; Burnout, Psychological | interventions — Sleep, REM; Amyloid

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, controlled and single-blind trial of 16 weeks. Students of Medicine, Nutrition, Psychology and Nursing are randomly assigned to the app group, the presential-based MBSR program or a waiting list. Three evaluations take place: pre-intervention, at 8 weeks (post-intervention) and at 16 weeks.
Who Masked: Outcomes Assessor
Masking Description: Single-blind. The type of intervention (presence-based, app or waiting list) can not be masked neither for the participant nor for the intervention provider. Thus, the masking only applies to the assessor of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: App. (Experimental): Participants use application "REM Volver a casa" on their cell phones during 8 weeks. Codes are provided to the students in order to unlock the different stages of the training free of charge. The application provides short videos and audios for training. Students practice on their own, in accordance with the instruction of completing a stage a week.
  Interventions: Behavioral: REM Volver a casa
- Group 2: MBSR. (Active Comparator): Participants attend a presence-based training during 8 weeks. The Mindfulness-Based Stress Reduction program involves a session of two and a half hours each week.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction program
- Group 3: Waiting list. (No Intervention): Participants do not receive any intervention during the study. At the end of the study (16 weeks), they are provided with the codes so they can unlock the app and use it like participants from Group 1.

INTERVENTIONS:
Behavioral: REM Volver a casa — The program aims to train the ability of the mind to focus attention on the present moment without judging, accepting the experience. REM is an application available for Android and iOs. It proposes a guided training through 8 stages. They contain video recordings with explanations about the fundamentals of mindfulness, audio recordings that guide practices of mindfulness, as well as suggestions to bring it into everyday life. They can be used whenever it suits the user. The app counts the progress of each participant, as well as the mood changes according to a distress scale before and after performing a formal practice. The app has been designed following the international recommendations for the development of apps (MARS guide).
  Other Names: REM, app
  Arms: Group 1: App.
Behavioral: Mindfulness-Based Stress Reduction program — The program aims to train the ability of the mind to focus attention on the present moment without judging, accepting the experience. MBSR is a program developed at the University of Massachusetts Medical Center in the 1970s by Professor Jon Kabat-Zinn. MBSR uses a combination of mindfulness meditation, body awareness, and yoga to help people become more mindful. In recent years, meditation has been the subject of clinical research, that suggests it may have beneficial effects, including stress reduction, relaxation, and improvements to quality of life. While MBSR has its roots in spiritual teachings, the program itself is secular. The session is delivered to a small group of people by a certified instructor during two and a half hours, every week.
  Other Names: MBSR
  Arms: Group 2: MBSR.

SUMMARY:
The main purpose of this study is to compare the efficacy of a mindfulness-based training app ('REM Volver a Casa') versus a regular, presence-based program (MBSR) on the reduction of anxiety and other factors related to the physician-patient relationship, in healthcare grade students.

DETAILED DESCRIPTION:
Healthcare students suffer from higher levels of anxiety and depression than the general population. It compromises not only their mental health, but also the quality of care provided. Aptitudes such as empathy and self-compassion are essential to improve this deficit and overcome the well-known burnout syndrome.

Mindfulness-Based Stress Reduction (MBSR) program has proven to be an effective intervention for lowering stress in numerous studies. However, this intervention asks for a significant degree of personal involvement, thus the number of dropouts is often reported as a problem. New technologies might allow users to adapt training to their personal schedules.

The present randomized trial aims to compare the efficacy of a mindfulness-based training delivered through a mobile application ('REM Volver a Casa'), a presence-based program (MBSR), and a control group in healthcare grade students.

ELIGIBILITY:
Inclusion Criteria:

* Student of Medicine, Nutrition, Psychology or Nursing.
* Ability to read and understand Spanish language.
* Signature of Informed Consent.

Exclusion Criteria:

* Previous MBSR or anorther standardized Mindfulness training.
* Inability to read or understand Spanish language.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
State-trait anxiety | From baseline to 8 weeks
  Post-intervention changes in State-Trait Anxiety Inventory (STAI) for each of the arms. It is a self-administered questionnaire which includes two subscales assessing state and trait anxiety. Each of them consists of 20 Likert items ranging 0-3. Lower values mean better outcomes.

SECONDARY OUTCOMES:
State-Trait Anger | From baseline to 8 weeks
  Post-intervention changes in State-Trait Anger Expression Inventory (STAXI) for each of the arms. It is a self-administered questionnaire that evaluates the experience, expression and control of anger, in adolescents and adults. The STAXI-2 Inventory consists of six scales and five subscales with 49 items in total.
Mindfulness | From baseline to 8 weeks
  Post-intervention changes in Five Facet Mindfulness Questionnaire (FFMQ) for each of the arms. FFMQ, by Baer, Smith, Hopkins, Krietemeyer and Toney (2006): 39 items that evaluate five facets on which the mindfulness ability is based: observe, describe, act with conscience, equanimity and not reactivity. Each item is scored according to a Likert scale that ranges from 1 (never) to 5 (very often). It has a high internal consistency, as well as a high predictive validity of the aspects that conform the Mindfulness construct (Baer, 2006). Validated in Spanish (Cebolla et al., 2012 ).
Self-compassion | From baseline to 8 weeks
  Post-intervention changes in dimensions of Neff Self-compassion Scale (SCS) for each of the arms. SCS (Neff, 2003), validated in Spanish in 2014 (García-Campayo et al., 2014 ): 26 items that evaluate six facets on which the self-compassion skill is based: kindness with oneself, judgment towards oneself, shared humanity, loneliness, mindfulness and overidentification. Each item is scored according to a Likert scale that ranges from 1 (almost never) to 5 (almost always).
Empathy | From baseline to 8 weeks
  Post-intervention changes in global Empathy questionnaire score (Jefferson Scale of Physician Empathy, JSE) for each of the arms. It includes three subscales: compassionate care, taking perspective and "standing on the patient's boots". Higher total values indicate greater empathy. It is valid in the Spanish population (Alcorta Garza et al., 2005).
Depression | From baseline to 8 weeks
  Post-intervention changes in Beck Depression Inventory (BDI-II) for each of the arms. Self-administered questionnaire of 21 items that measures the severity of depression in adults and adolescents over 13 years of age. It is one of the most used questionnaires within the field of psychology when measuring the severity of depression.
Expectancy of improvement | Pre-intervention questionnaire
  Pre-intervention measure through the 0-100% Expectancy of Improvement Scale, derived from Credibility / Expectancy Questionnaire (CEQ, Devilly & Borkovec), which has proven to be a reliable predictor of results in multiple studies and populations. The CEQ questionnaire is the measure of credibility / expectations most used in research in psychotherapy. The scale is graduated in 10 options, corresponding higher score to greater expectation of improvement.
Autonomous motivation | Pre-intervention questionnaire
  Pre-intervention measure through the Self-Regulation Questionnaire (SRQ-L, Williams, GC, & Deci, 2000). It is given a version of this self-administered questionnaire, which provides subscales of autonomous, controlled motivation and an autonomous regulation index (RAI, which is the subtraction of the previous). It has been previously used in medical students showing evidence of criterion validity with other measures. The questionnaire includes 13 reasons for participation in the intervention, in which the participant must score from 0 to 7 on a Likert scale if each statement is true for their case.
State-Trait Anxiety | From baseline to 16 weeks
  Post-intervention changes in State-Trait Anxiety Inventory (STAI) for each of the arms. It is a self-administered questionnaire which includes two subscales assessing state and trait anxiety. Each of them consists of 20 Likert items ranging 0-3. Lower values mean better outcomes.
Mindfulness | From baseline to 16 weeks
  Post-intervention changes in Five Facet Mindfulness Questionnaire (FFMQ) for each of the arms. FFMQ, by Baer, Smith, Hopkins, Krietemeyer and Toney (2006): 39 items that evaluate five facets on which the mindfulness ability is based: observe, describe, act with conscience, equanimity and not reactivity. Each item is scored according to a Likert scale that ranges from 1 (never) to 5 (very often). It has a high internal consistency, as well as a high predictive validity of the aspects that conform the Mindfulness construct (Baer, 2006). Validated in Spanish (Cebolla et al., 2012 ).
State-Trait Anger | From baseline to 16 weeks
  Post-intervention changes in State-Trait Anger Expression Inventory (STAXI) for each of the arms. It is a self-administered questionnaire that evaluates the experience, expression and control of anger, in adolescents and adults. The STAXI-2 Inventory consists of six scales and five subscales with 49 items in total.
Self-compassion | From baseline to 16 weeks
  Post-intervention changes in dimensions of Neff Self-compassion Scale (SCS) for each of the arms. SCS (Neff, 2003), validated in Spanish in 2014 (García-Campayo et al., 2014 ): 26 items that evaluate six facets on which the self-compassion skill is based: kindness with oneself, judgment towards oneself, shared humanity, loneliness, mindfulness and overidentification. Each item is scored according to a Likert scale that ranges from 1 (almost never) to 5 (almost always).
Empathy | From baseline to 16 weeks
  Post-intervention changes in global Empathy questionnaire score (Jefferson Scale of Physician Empathy, JSE) for each of the arms. It includes three subscales: compassionate care, taking perspective and "standing on the patient's boots". Higher total values indicate greater empathy. It is valid in the Spanish population (Alcorta Garza et al., 2005).
Depression | From baseline to 16 weeks
  Post-intervention changes in Beck Depression Inventory (BDI-II) for each of the arms. Self-administered questionnaire of 21 items that measures the severity of depression in adults and adolescents over 13 years of age. It is one of the most used questionnaires within the field of psychology when measuring the severity of depression.

OTHER OUTCOMES:
Practice time | 8 weeks
  In Group 1, practice time is measured by the app. In Group 2, participants are asked to note down practice time.
Drop-out rate | From baseline to 8 weeks
  Drop-out rate during the study in each arm.
Drop-out rate | From baseline to 16 weeks
  Drop-out rate during the study in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Bayón, Doctor, Principal Investigator — Hospital Universitario La Paz. Universidad Autónoma de Madrid; Beatriz Rodríguez Vega, Doctor, Principal Investigator — Hospital Universitario La Paz. Universidad Autónoma de Madrid
Locations (1):
- Hospital Universitario La Paz [La Paz University Hospital], Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared from PI on request

REFERENCES:
- [Background] Aherne D, Farrant K, Hickey L, Hickey E, McGrath L, McGrath D. Mindfulness based stress reduction for medical students: optimising student satisfaction and engagement. BMC Med Educ. 2016 Aug 18;16(1):209. doi: 10.1186/s12909-016-0728-8. PMID 27535243
- [Background] Barbosa P, Raymond G, Zlotnick C, Wilk J, Toomey R 3rd, Mitchell J 3rd. Mindfulness-based stress reduction training is associated with greater empathy and reduced anxiety for graduate healthcare students. Educ Health (Abingdon). 2013 Jan-Apr;26(1):9-14. doi: 10.4103/1357-6283.112794. PMID 23823667
- [Background] Krusche A, Cyhlarova E, Williams JM. Mindfulness online: an evaluation of the feasibility of a web-based mindfulness course for stress, anxiety and depression. BMJ Open. 2013 Nov 29;3(11):e003498. doi: 10.1136/bmjopen-2013-003498. PMID 24293203
- [Background] Lamothe M, Rondeau E, Malboeuf-Hurtubise C, Duval M, Sultan S. Outcomes of MBSR or MBSR-based interventions in health care providers: A systematic review with a focus on empathy and emotional competencies. Complement Ther Med. 2016 Feb;24:19-28. doi: 10.1016/j.ctim.2015.11.001. Epub 2015 Nov 27. PMID 26860797
- [Background] Kirby JN. Compassion interventions: The programmes, the evidence, and implications for research and practice. Psychol Psychother. 2017 Sep;90(3):432-455. doi: 10.1111/papt.12104. Epub 2016 Sep 24. PMID 27664071
- See also: App webpage — http://remvolveracasa.com/